CLINICAL TRIAL: NCT00000428
Title: Combining N-of-1 Trials to Assess Fibromyalgia Therapies
Brief Title: Combining N-of-1 Trials to Assess Fibromyalgia Treatments
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tufts Medical Center (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Deborah Zucker, MD, PhD, Tufts-New England Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01AR045416 (NIH); R01AR045416 (NIH); NIAMS-038
Record Dates: First submitted 2000-01-18; First posted 2000-01-19 (Estimated); Last update posted 2013-08-01 (Estimated); Status verified 2013-07

CONDITIONS: Fibromyalgia
Keywords: Fibromyalgia Syndrome (FMS); Amitriptyline; Fluoxetine
MeSH Terms: conditions — Fibromyalgia | interventions — Amitriptyline; Fluoxetine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): Patients received each intervention multiple times in random-order crossover design.
  Interventions: Drug: Amitriptyline; Drug: Amitriptyline plus Fluoxitine

INTERVENTIONS:
Drug: Amitriptyline — Amitriptyline 25 mg po
  Other Names: Elavil
Drug: Amitriptyline plus Fluoxitine — Amitriptyline 25 mg po plus Fluoxitine 20 mg po
  Other Names: elavil plus prozac

SUMMARY:
This study will compare the effectiveness of combination therapy with the drugs amitriptyline and fluoxetine (AM+FL) and amitriptyline (AM) alone in the treatment of people with fibromyalgia. Doctors will treat each study participant with both AM + FL and AM alone for 6 weeks at a time. The study uses a method that combines results from treatment of individual patients to assess overall treatment effectiveness and help individual patients and their physicians with their treatment decisions. This study will also help compare the results of community-based studies (studies involving private doctors) and studies based at clinical research centers.

DETAILED DESCRIPTION:
This study will use the combined N-of-1 method to compare the effectiveness of the combination therapy amitriptyline and fluoxetine (AM+FL) versus amitriptyline (AM) alone in patients with fibromyalgia (FM). It will also compare community-based and center-based trial results. We will ask community-based, board-certified rheumatologists to participate as investigators and we will also carry out a center-based study (at Newton-Wellesley Hospital). Physicians will ask patients meeting eligibility criteria to participate in this study and undergo an N-of-1 trial.

Each N-of-1 trial will consist of three paired crossover periods (each 6-weeks long) during which the patient will receive either AM + placebo (placebo every morning and AM 25 mg at night) or combination treatment AM+FL (FL 20 mg in the morning and AM 25 mg at night). The dispensing pharmacy will carry out paired randomization.

We will assess patient evaluations and outcome measures at baseline prior to trial, at the end of each treatment period, and 3 months after completion of the N-of-1 trial. In addition, at baseline, we will obtain demographic information, an electrocardiogram, and baseline blood tests. We may ask patients to have additional blood tests at the period evaluations. We will also do a pregnancy test for all women of child-bearing age enrolling in the study. The main study outcome measure will be the Fibromyalgia Impact Questionnaire (FIQ). Additional measures will include the Visual Analog Scales (VAS) for pain, sleep, global well-being; Physician VAS for global well-being; and tender-point score.

We will analyze the results of the N-of-1 trials in two ways: (1) using only the individual patient's results (classic one-sided t-test) and (2) using the patient's results in combination with the results of other patients who underwent similar trials (the combined N-of-1 approach). To obtain the latter information, we will include each patient's results for the collective analysis. We will provide these results back to the physicians and will record the final treatment decisions the physicians reach with their patients. In addition, we will ask both physicians and patients to comment on their participation in an N-of-1 trial and this research process. Followup of patients 3 months after completion of their N-of-1 trial will include determining current medication and a current outcome assessment. Investigators will record all adverse drug reactions and patients withdrawn from studies. They will also record the reason for withdrawal for all patients choosing to withdraw. We will include results from patients who drop out due to reasons other than drug reactions in the combined N-of-1 analyses if completed period pair results are available. An independent safety officer will review all withdrawals.

Results of individual patient trials will be confidential; however, we will combine these results (after removal of patient identifiers) with the results of other patients, and will publish the overall results of this study. We will maintain the connection of results to patient identifiers only to enable us to provide results to individual investigators and their patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet fibromyalgia criteria as defined by the American College of Rheumatology
* No systemic illness (current or past) or other contraindications to taking study medications (e.g. known hypersensitivity)
* Age 18-60
* Patient willingness, and physician agreement, to discontinue CNS medications/NSAIDs/analgesics for 1 week prior to starting their trial
* Patient informed consent and agreement to participate in an N-of-1 trial

Exclusion Criteria:

* Patients who are currently pregnant or who plan to become pregnant during the study period
* Patients with any contraindications to using either amitriptyline or fluoxetine

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 58 (Actual)
Dates: Start 2000-09; Primary Completion 2004-03 (Actual); Study Completion 2004-03 (Actual)

PRIMARY OUTCOMES:
FIbromyalgia Impact Questionnaire scores | At baseline,each treatment period, and at 3 mo follow up

CONTACTS AND LOCATIONS:
Overall Officials: Deborah R. Zucker, Principal Investigator — New England Medical Center, Tufts University School of Medicine
Locations (7):
- United States (7):
  - Office of Raphael Kieval, MD, Brockton, Massachusetts
  - Office of Ronald J. Rapoport, MD, Fall River, Massachusetts
  - Office of Eileen Winston, MD, Framingham, Massachusetts
  - Office of Nicola Mogavero, MD, Melrose, Massachusetts
  - Office of Jacqueline Feuer, MD, Needham, Massachusetts
  - Newton-Wellesley Hospital, Newton, Massachusetts
  - Office of Sharon A. Stotsky, MD, North Reading, Massachusetts

REFERENCES:
- [Background] Goldenberg D, Mayskiy M, Mossey C, Ruthazer R, Schmid C. A randomized, double-blind crossover trial of fluoxetine and amitriptyline in the treatment of fibromyalgia. Arthritis Rheum. 1996 Nov;39(11):1852-9. doi: 10.1002/art.1780391111. PMID 8912507
- [Background] Zucker DR, Schmid CH, McIntosh MW, D'Agostino RB, Selker HP, Lau J. Combining single patient (N-of-1) trials to estimate population treatment effects and to evaluate individual patient responses to treatment. J Clin Epidemiol. 1997 Apr;50(4):401-10. doi: 10.1016/s0895-4356(96)00429-5. PMID 9179098
- [Background] Guyatt G, Sackett D, Taylor DW, Chong J, Roberts R, Pugsley S. Determining optimal therapy--randomized trials in individual patients. N Engl J Med. 1986 Apr 3;314(14):889-92. doi: 10.1056/NEJM198604033141406. PMID 2936958
- [Background] Guyatt G, Sackett D, Adachi J, Roberts R, Chong J, Rosenbloom D, Keller J. A clinician's guide for conducting randomized trials in individual patients. CMAJ. 1988 Sep 15;139(6):497-503. PMID 3409138
- [Background] Larson EB. N-of-1 clinical trials. A technique for improving medical therapeutics. West J Med. 1990 Jan;152(1):52-6. PMID 2309473
- [Result] Zucker DR, Ruthazer R, Schmid CH, Feuer JM, Fischer PA, Kieval RI, Mogavero N, Rapoport RJ, Selker HP, Stotsky SA, Winston E, Goldenberg DL. Lessons learned combining N-of-1 trials to assess fibromyalgia therapies. J Rheumatol. 2006 Oct;33(10):2069-77. PMID 17014022